CLINICAL TRIAL: NCT00111267
Title: The Effect of Oral Vitamin B12 Supplementation on Cognitive Performance in Elderly People: the Brain12 Study
Brief Title: Oral Vitamin B12 Supplementation and Cognitive Performance in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P03.0277L; ZonMW 2100.0067
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Cognitive Decline; Cognitive Symptoms
Keywords: vitamin B12; cognitive function; oral supplementation; elderly
MeSH Terms: conditions — Cognitive Dysfunction; Neurobehavioral Manifestations | interventions — Vitamin B 12

INTERVENTIONS:
Behavioral: vitamin B12 supplementation
Behavioral: vitamin B12 + folic acid combined supplementation

SUMMARY:
The purpose of this trial is to study the effects of oral vitamin B12 supplementation and vitamin B12 combined with folic acid supplementation on cognitive performance for 24 weeks in elderly people with mild vitamin B12 deficiency.

DETAILED DESCRIPTION:
Mild vitamin B12 deficiency is highly prevalent in old age. Reasons for this high prevalence are not fully understood, but include atrophic gastritis and bacterial overgrowth which affect the absorption (active) of food-bound vitamin B12. In contrast, the ability to absorb crystalline vitamin B12 (e.g. the form found in fortified foods or vitamin pills) remains intact in old age. In both healthy and cognitively impaired elderly people, associations between vitamin B12 status and cognitive performance have been observed, and the follow-up of geriatric patients suggests effects of parenteral treatment in early cognitive impairment.

We investigated whether daily oral supplementation with 1,000 μg vitamin B12 or 1,000 μg vitamin B12 combined with 400 μg folate for 24 weeks improves cognitive performance in people over 70 years with vitamin B12 deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Mild vitamin B12 deficiency:

  * Low plasma vitamin B12 concentration (100 < B12 < 300 pmol/L)
  * Elevated methylmalonic acid (MMA) concentration (> 0.32 umol/L)
  * Creatinine concentration < 120 umol/L

Exclusion Criteria:

* Severe cognitive impairment
* Anemia
* Gastrointestinal surgery or diseases
* Use of vitamin B12 injections or supplements containing > 25 ug vitamin B12 and/or 200 ug folic acid
* < 90% compliance during a 2 week placebo run in period
* No written informed consent
* Participation in other research studies

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 165
Dates: Start 2003-05; Study Completion 2005-01

PRIMARY OUTCOMES:
Cognitive performance in the domains of attention, concentration, memory, executive function, speed

SECONDARY OUTCOMES:
Blood biochemistry including vitamin B12, methylmalonic acid, holotranscobalamin, homocysteine, and red blood cell folate

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands